CLINICAL TRIAL: NCT03509714
Title: Oxaloacetate Supplementation for Emotional PMS; Measuring Improvements in Depression, Anxiety, Perceived Stress, and Aggression
Brief Title: Oxaloacetate Supplementation for Emotional PMS
Acronym: OAA4PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terra Biological LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EmotionalPMS1; TV-OX-108 (Other: The Institute for Regenerative and Cellular Medicine)
Record Dates: First submitted 2018-04-06; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Premenstrual Syndrome (PMS)
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Baseline measurement of all participants. Randomized double-blinded placebo controlled crossover study for Phase 1. Due to carry-over effects, Phase 2 of the study started each participant with placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Oxaloacetate/Vitamin C capsules were bottled in 30 count HDPE bottles. Placebo capsules (rice flour) were manufactured to similar size capsules and bottles. Bottles were labeled either Group A or Group 1. Code was broken at the end of Phase 1 of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Part 1 Oxaloacetate Random (Active Comparator): Participants take 2 capsules Jubilance 100 mg Oxaloacetate/150 mg Ascorbic Acid blend per day during their entire menstrual cycle (approximately 28 days) or 2 capsules of 250 mg rice flour (Placebo). After one menstrual cycle, they cross-over to the other option.
  Interventions: Dietary Supplement: Jubilance (100 mg Oxaloacetate/150 mg Ascorbic Acid); Dietary Supplement: rice flour (Placebo)
- Experimental: Part 2 Oxaloacetate Second (Active Comparator): Participants take 2 capsules of 250 mg rice flour (Placebo) per day during their entire menstrual cycle (approximately 28 days). After one menstrual cycle, they cross-over to 2 capsules of Jubilance 100 mg Oxaloacetate/150 mg Ascorbic Acid blend.
  Interventions: Dietary Supplement: Jubilance (100 mg Oxaloacetate/150 mg Ascorbic Acid); Dietary Supplement: rice flour (Placebo)

INTERVENTIONS:
Dietary Supplement: Jubilance (100 mg Oxaloacetate/150 mg Ascorbic Acid) — 2 Pills to be taken orally per day during their entire menstrual cycle
  Other Names: Jubilance for Emotional PMS
Dietary Supplement: rice flour (Placebo) — 250 mg rice flour (Placebo)

SUMMARY:
Emotional Premenstrual Syndrome (PMS) affects millions of women worldwide. For Emotional PMS, including depression, anxiety, perceived stress and aggression, there are very few options. Recent observational data suggest that nutritional supplementation with oxaloacetate, a human energy metabolite, greatly reduced the symptoms of Emotional PMS. The aim of this study was to confirm these observations on the effects of oxaloacetate on Emotional PMS symptom severity within a controlled clinical trial setting.

DETAILED DESCRIPTION:
Oxaloacetate is an energy metabolite found in every cell of the human body. It holds a key place in the Krebs Cycle within the mitochondria, providing energy to the cells. It is also a critical early metabolite in gluconeogenesis, which provides glucose for the heart and brain during times of low glucose. It is critical to human metabolism, proper cellular function and it is central to energy production and use in the body.

Oxaloacetate may affect Emotional PMS through multiple mechanisms. During PMS, there is a large increase in glucose utilization in the cerebellum of the brain in women who are affected with emotional mood swings. Oxaloacetate supplementation has been shown to support proper glucose levels in the body. Having an excess of oxaloacetate allows gluconeogenesis take place upon demand, thereby fueling the brain, and perhaps meeting cerebellum glucose need.

In addition to oxaloacetate's ability to support proper glucose regulation, oxaloacetate affects two chemicals in the brain, GABA and glutamate. Altering the GABA/Glutamate ratio can affect mood. Oxaloacetate supplementation can reduce glutamate levels in the brain via a process called "Glutamate Scavenging". In addition, oxaloacetate supplementation was shown to increase GABA levels in animal models. By both lowering glutamate and increasing GABA, the GABA/Glutamate ratio is affected, which may also help women with Emotional PMS.

This study will investigate oxaloacetate's effect on Emotional PMS using patient completed surveys to measure depression, anxiety, perceived stress, and aggression, and statistically compare these results against placebo (rice flour) and baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* Women with Emotional Premenstrual Syndrome (PMS),
* Women who speak English as their primary language
* Women who understand the Human Consent Form
* Ability to swallow capsules

Exclusion Criteria:

* Formal diagnosis of clinical depression
* Formal diagnosis of premenstrual dysphoric disorder (PMDD).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Depression associated with Emotional PMS | Change from baseline value to value after supplementation for entire menstrual cycle (about 28 days) for each study arm in cross-over design (3 data points compared 1 at baseline 1 after menstrual cycle 1 and 1 after menstrual cycle 2).
  Depression as measured during Emotional PMS with Beck's Depression Inventory Survey, which scores depression with 26 questions rated 0 to 3. Total score ranges from 0 to 78. Higher values indicate worse depression.
Anxiety associated with Emotional PMS | Change from baseline value to value after supplementation for one entire menstrual cycle (about 28 days) for each study arm in cross-over design (3 data points compared 1 at baseline 1 after menstrual cycle 1 and 1 after menstrual cycle 2).
  Anxiety as measured during Emotional PMS with Generalized Anxiety Disorder Survey, which scores anxiety with 7 questions rated 0 to 3. Total score ranges from 0 to 21. Higher values indicate worse anxiety.
Perceived Stress with Emotional PMS | Change from baseline value to value after supplementation for one entire menstrual cycle (about 28 days) for each study arm in cross-over design (3 data points compared 1 at baseline 1 after menstrual cycle 1 and 1 after menstrual cycle 2).
  Perceived Stress as measured during Emotional PMS with Cohen's Perceived Stress Survey, which scores perceived stress with 9 questions rated 0 to 4. Total score ranges from 0 to 36. Higher values indicate worse perceived stress.
Aggression with Emotional PMS | Change from baseline value to value after supplementation for one entire menstrual cycle (about 28 days) for each study arm in cross-over design (3 data points compared 1 at baseline 1 after menstrual cycle 1 and 1 after menstrual cycle 2).
  Aggression as measured during Emotional PMS with Buss-Perry Aggression Scale, which scores depression with 29 questions rated 1 to 5. Total score ranges from 29 to 145. Higher values indicate worse aggression.
Adverse Event Reporting | Through study completion, an average of 60 days (2 menstrual cycles)
  Safety of oxaloacetate supplementation in Emotional PMS patients

SECONDARY OUTCOMES:
Suicidal Ideation with Emotional PMS | Change from baseline value to value after supplementation for one entire menstrual cycle (about 28 days) for each study arm in cross-over design (3 data points compared 1 at baseline 1 after menstrual cycle 1 and 1 after menstrual cycle 2).
  Suicidal Ideation as measured with a subscale of Beck's Depression Inventory, with a scale ranging from 0 to 3 in women who initially record suicidal ideation of greater than 0.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Tully, PhD, Study Director — Energy Medicine research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams DS, Cash A, Hamadani L, Diemer T. Oxaloacetate supplementation increases lifespan in Caenorhabditis elegans through an AMPK/FOXO-dependent pathway. Aging Cell. 2009 Dec;8(6):765-8. doi: 10.1111/j.1474-9726.2009.00527.x. Epub 2009 Sep 30. PMID 19793063
- [Background] Yoshikawa K. Studies on the anti-diabetic effect of sodium oxaloacetate. Tohoku J Exp Med. 1968 Oct;96(2):127-41. doi: 10.1620/tjem.96.127. No abstract available. PMID 4884771
- [Background] Rapkin AJ, Berman SM, Mandelkern MA, Silverman DH, Morgan M, London ED. Neuroimaging evidence of cerebellar involvement in premenstrual dysphoric disorder. Biol Psychiatry. 2011 Feb 15;69(4):374-80. doi: 10.1016/j.biopsych.2010.09.029. Epub 2010 Nov 18. PMID 21092938
- [Background] Schmahmann JD. The role of the cerebellum in cognition and emotion: personal reflections since 1982 on the dysmetria of thought hypothesis, and its historical evolution from theory to therapy. Neuropsychol Rev. 2010 Sep;20(3):236-60. doi: 10.1007/s11065-010-9142-x. Epub 2010 Sep 7. PMID 20821056
- [Background] Wilkins HM, Harris JL, Carl SM, E L, Lu J, Eva Selfridge J, Roy N, Hutfles L, Koppel S, Morris J, Burns JM, Michaelis ML, Michaelis EK, Brooks WM, Swerdlow RH. Oxaloacetate activates brain mitochondrial biogenesis, enhances the insulin pathway, reduces inflammation and stimulates neurogenesis. Hum Mol Genet. 2014 Dec 15;23(24):6528-41. doi: 10.1093/hmg/ddu371. Epub 2014 Jul 15. PMID 25027327
- [Derived] Tully L, Humiston J, Cash A. Oxaloacetate reduces emotional symptoms in premenstrual syndrome (PMS): results of a placebo-controlled, cross-over clinical trial. Obstet Gynecol Sci. 2020 Mar;63(2):195-204. doi: 10.5468/ogs.2020.63.2.195. Epub 2020 Feb 25. PMID 32206660